CLINICAL TRIAL: NCT03240887
Title: The Evaluation of Peer Group Connection in Rural North Carolina and New York City, New York
Brief Title: Evaluation of Peer Group Connection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Policy & Research Group (Other)
Collaborators: The Office of Adolescent Health, HHS (U.S. Federal Agency); Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6 TP2AH000037-01-01
Record Dates: First submitted 2017-07-27; First posted 2017-08-07 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Pregnancy in Adolescence
Keywords: Teen pregnancy prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Group Connection (PGC) (Experimental): Ninth-grade participants are assigned to small groups of 10-14 students that attend weekly peer group outreach sessions led by older peer leaders.
  Interventions: Behavioral: Peer Group Connection
- Business as usual (No Intervention): Ninth grade students remain in their regularly scheduled school classes or activities during PGC outreach times.

INTERVENTIONS:
Behavioral: Peer Group Connection — Faculty advisors at each participating high school are trained to run the program and teach a daily leadership course to peer leaders. Eleventh and twelfth-grade peer leaders who participate in the daily leadership development class facilitate outreach sessions with their assigned group of ninth graders. PGC can be offered in either a half-year (semester) or full-year format. In either format, a minimum of 18, 45-minute outreach sessions are expected to be offered to PGC participants during the course of their ninth-grade year. Outreaches are created to facilitate the transition to high school and encourage students to attend school, set goals for themselves, and make healthy decisions.
  Arms: Peer Group Connection (PGC)

SUMMARY:
A randomized controlled trial is being conducted in high schools in North Carolina and New York City to determine the impact of a school-based, positive youth development program on sexual behaviors associated with teen pregnancy

DETAILED DESCRIPTION:
The Policy & Research Group (PRG) is conducting a rigorous evaluation of the Peer Group Connection (PGC) program's impact on sexual behaviors associated with teen pregnancy. PGC is a school-based, group peer mentoring program for ninth grade students that is designed to facilitate the transition into high school and improve non-cognitive abilities, student engagement, and educational outcomes. The study enrolls students from high schools that serve large populations of economically disadvantaged and minority students in communities with high teenage birth rates. In North Carolina, the study is being implemented in schools serving rural populations, and in New York City, schools serving largely Hispanic and other minority populations are targeted.

As part of the PGC program, ninth-grade participants attend weekly group outreach sessions led by older peer leaders. Outreach sessions occur during regularly scheduled classes (participants are pulled from their classes to attend). They include hands-on activities, simulations, and discussions intended to build group cohesion and to improve the decision-making skills of group members. A minimum of 18, 45-minute outreach sessions are expected to be offered to PGC participants during the course of their ninth-grade year. Although PGC is not explicitly a sexual health or teen pregnancy prevention program, the belief is that by engaging ninth grade students in school, building connectedness among peers, and building students' decision-making and goal-setting skills, PGC will encourage students to make healthier decisions, including reducing sexual risk-taking and increasing protective behaviors.

The comparison condition consists of normally scheduled classes or activities (e.g., Physical Education/Health class, elective class, or homeroom period) that comparison group participants are assigned to during the period that PGC outreaches occur. Comparison group participants will therefore receive more time in the regularly scheduled class than will the treatment group, but there will be no alternative program or additional activities offered to the participants assigned to the comparison group.

The study is an individual randomized controlled trial in which eligible, consenting ninth grade participants are randomly assigned by the evaluator to intervention (PGC) or control (class as usual) groups at a 1:1 ratio. Outcomes will be assessed using questionnaire data gathered at three time points: baseline, occurring during the fall of participants' 9th grade year (prior to the provision of any PGC programming), and follow-up during the fall of their 10th and 11th grade years. Primary outcomes of interest include sexual initiation, frequency of any type of sex, and number of sexual partners.

ELIGIBILITY:
Inclusion Criteria:

1. Be enrolled at a study school
2. Provide parental consent and personal assent to participate in the study
3. Meet basic requirements for data collection (students must have the ability to complete a self-administered Participant Questionnaire, which is available in English and Spanish, in a classroom or group setting, unassisted, in 60 minutes or less.)
4. Be entering the ninth grade for the first time.

Exclusion Criteria:

1. Be intending to enroll in a non-study school in ninth grade.
2. Be repeating ninth grade.
3. Be unable to complete the questionnaire without assistance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1523 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Sexual initiation | 1 year after baseline, or the beginning of the 10th grade
  The measure is operationalized as a dichotomous outcome, where 1 = participant has had sex, 0 = participant has never had sex. One questionnaire item measures sexual initiation: Have you ever had any type of sex (oral, vaginal, or anal)?
Frequency of sex | 1 year after baseline, or the beginning of the 10th grade
  The outcome is operationalized as the count of the number of times a participant reports having had any type of sex in the past 3 months. One questionnaire item measures frequency of sex: In the past 3 months, how many times have you had any type of sex?
Number of sexual partners | 1 year after baseline, or the beginning of the 10th grade
  The outcome is operationalized as the count of the number of sexual partners a participant reports having in the past 3 months. Two questionnaire items are used to measure the number of sexual partners questions. The first item asks the participant with whom they have had sexual contact during their life, and if sexual contact with any gender is reported, the second item subsequently asks how many sexual partners they have had in the past three months.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jenner, Ph.D., Principal Investigator — The Policy & Research Group
Locations (1):
- The Policy & Research Group, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A dataset will be prepared at the conclusion of the study, which includes de-identified individual-level data on all study participants who contributed self-report data. Respondents will be represented only by a research ID number. Included in the dataset will be self-report data collected across all survey administrations (including demographic characteristics, sexual behaviors, and theoretical antecedents to those behaviors) and select information on program participation (e.g., which program sessions were attended). Basic data cleaning steps will be taken in order to ensure data are unidentifiable and to increase usability.
Time Frame: The individual participant dataset will become available twelve months after the study has concluded.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT03240887/Prot_SAP_001.pdf